CLINICAL TRIAL: NCT01129661
Title: An Adaptive, Phase I, Single-Centre, Randomised, Double-blind, Placebo-controlled Single Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics, of Intravenous CSL112 in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of CSL112 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSLCT-HDL-09-63
Record Dates: First submitted 2010-05-19; First posted 2010-05-25 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
MeSH Terms: interventions — CSL112; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (0.9%) (Placebo Comparator)
  Interventions: Biological: normal saline (0.9%)
- CSL112 (Experimental)
  Interventions: Biological: CSL112 (reconstituted HDL)

INTERVENTIONS:
Biological: CSL112 (reconstituted HDL) — Single escalating intravenous doses of CSL112
  Arms: CSL112
Biological: normal saline (0.9%) — Single intravenous dose of normal saline (0.9%)
  Arms: normal saline (0.9%)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of escalating doses of CSL112 after single intravenous infusions in healthy volunteers and to measure the pharmacokinetics of CSL112 after single intravenous infusions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 18 years to less than 55 years
* Body weigh 45 kg or greater

Exclusion Criteria:

* Evidence of a clinically significant medical condition, disorder or disease
* Evidence of clinically relevant abnormal laboratory test result
* Evidence of history of alcohol or substance abuse

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by the frequency of drug-related clinical adverse events. | Up to 14 days after infusion of CSL112
Safety and tolerability as measured by liver function tests. | Up to 14 days after infusion of CSL112

SECONDARY OUTCOMES:
Pharmacokinetics of lipoprotein. | Up to 10 days after infusion of CSL112
  Plasma levels of lipoprotein.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Zheng B, Duffy D, Tricoci P, Kastrissios H, Pfister M, Wright SD, Gille A, Tortorici MA. Pharmacometric analyses to characterize the effect of CSL112 on apolipoprotein A-I and cholesterol efflux capacity in acute myocardial infarction patients. Br J Clin Pharmacol. 2021 Jun;87(6):2558-2571. doi: 10.1111/bcp.14666. Epub 2020 Dec 23. PMID 33217027